CLINICAL TRIAL: NCT06618677
Title: Efficacy of a Low FODMAP Diet in IBS Children and Impact on Microbiota, Urinary and Faecal Metabolome
Brief Title: Efficacy of a Low FODMAP Diet in IBS Children and Impact on Urinary and Faecal Metabolome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Prof, University of Bari
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IBS-FODMAP
Record Dates: First submitted 2023-04-24; First posted 2024-10-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: IBS; Functional Gastrointestinal Disorders
Keywords: FODMAPs; IBS
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — FODMAP Diet

STUDY DESIGN:
Intervention Model Description: single center, prospective, single blind low versus standard FODMAPs diet trial with crossover
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LOW FODMAP-wash out- STANDARD FODMAPs (Active Comparator): Arm starting with low fodmap diet
  Interventions: Other: LOW FODMAPs Diet
- STANDARD FODMAPs-wash out-LOW FODMAP (Active Comparator): Arm starting with standard fodmap diet
  Interventions: Other: LOW FODMAPs Diet

INTERVENTIONS:
Other: LOW FODMAPs Diet — patients will be randomized to low or standard FODMAP diet for 14 days; then, children from both arms started the wash-out period of two weeks and subsequently started the final 2-week period on standard or low FODMAP diet. The LFD will have a FODMAP content expressed in grams 0.15 g/kg/d FODMAPs (maximum 10 g/day) while the SFD will contain 0.7 g/kg/d FODMAPs (maximum 60 g/day).
  Other Names: STANDARD FODMAPs Diet

SUMMARY:
Irritable bowel syndrome (IBS) is a functional gastrointestinal disorder characterized by abdominal pain associated with defecation, or changes in stool frequency or stool form .

The low FODMAPs diet (LFD) is a relatively new approach in the management of IBS and focuses on limiting intake of poorly absorbed carbohydrates.

FODMAPs are highly fermentable but poorly absorbed short-chain carbohydrates and polyols contained in a wide variety of foods. FODMAPs include oligosaccharides (fructans, fructo-oligosaccharides = FOS and galacto-oligosaccharides = GOS), disaccharides (lactose), monosaccharides (fructose), and polyols (sorbitol, mannitol, maltitol, xylitol, polydextrose, and isomalt).

Many studies and meta-analysis in adults have shown that a low FODMAPs diet is effective in reducing IBS symptoms, particularly bloating and abdominal pain. On the other hand, evidences in children are scarce.

Previous studies in adults have demonstrated differences in urine metabolites between IBS patients receiving LFD compared to a high FODMAP diet (HFD), providing interesting hypotheses for pathophysiological mechanisms in IBS.

Aim of this study is to evaluate the efficacy of a LFD on gastrointestinal symptoms in children with IBS. Moreover, the investigators will assess the impact of LFD vs a diet with a standard content of FODMAPs (SFD) on the fecal and urinary metabolomic profile of pediatric IBS patients.

This is a single center, prospective, single blind low versus standard FODMAPs diet trial with crossover performed at Pediatric Gastroenterology Unit at the University of Bari.

The trial includes four phases (run-in, low FODMAP diet, wash out and standard FODMAP diet). The run-in phase (weeks 1-2) aim to assess basal symptoms while on habitual diet and only symptomatic children (VAS>3) will progress to the dietetic intervention trial.

Then patients will be randomized to low or standard FODMAP diet for 14 days; then, children from both arms start the wash-out period of two weeks and subsequently start the final 2-week period on standard or low FODMAP diet.

DETAILED DESCRIPTION:
Single center, prospective, single blind low versus standard FODMAPs diet trial with crossover performed at Pediatric Gastroenterology Unit at the University of Bari Metabolomic analysis will be performed at Department of Soil, Plant and Food Science, University of Bari Aldo Moro.

The study will include all consecutive patients diagnosed with IBS according to the Rome IV criteria at Giovanni XXII Children's Hospital of Bari. The Giovanni XXII Children's Hospital of Bari is the tertiary referral center for the diagnosis and follow-up of gastrointestinal disorders in our region, covering an estimated population of 1400000 children, (National Institute of Statistics-https://www.istat.it accessed on 1 January 2023) with more than 10000 children followed up in the gastrointestinal clinic.

The trial includes four phases (run-in, low FODMAP diet, wash out and standard FODMAP diet). The run-in phase (weeks 1-2) aim to assess basal symptoms while on habitual diet and only symptomatic children (VAS>3) will progress to the dietetic intervention trial.

Then patients will be randomized to low or standard FODMAP diet for 14 days; then, children from both arms start the wash-out period of two weeks and subsequently start the final 2-week period on standard or low FODMAP diet. The order of the dietetic regimens is established according a computer-generated randomization list.

Fecal and urinary samples for analyzing metabolome will be collected before interventions and at the end of each dietetic regimen.

The study adheres to the Declaration of Helsinki, was approved by the institutional ethical committee. All patients gave full written informed consent.

Dietetic intervention An experienced dietician will design two different dietetic regimens (SFD and LFD), as a tailored personalized menu of 2 weeks duration, with manual calculation of nutrients and kilocalories according child age and weight. At enrollment the dietician will explain the diets in detail to the families who will be not aware of the content of FODMAP (low vs. standard). Parents will be only advised that the purpose of the study is to "Assess whether changing the amount of certain foods in the diet could affects symptoms of IBS" and the concept of FODMAPs wont be never mentioned during the study. Both menus will be normocaloric and balanced in macro- and micronutrients in relation to the age of the patient under study, according to the main principles of the Mediterranean diet. All menus comprise five meals during the day: breakfast, snack, lunch, snack and dinner. Food options present in the menus will be agree between the dietician, parents and children.

The food intake will be recorded on a diary and the same dietician, during follow-up visits checked dietary compliance. A proper dietary adherence was defined if percentage of amount of food left was less than 10% and number of times non-compliant per week was less than 2.

ELIGIBILITY:
Inclusion Criteria:

a) age between 4 and 18 years; b) diagnosis of IBS according to Rome IV criteria; c) absence of other organic diseases; d) feeding via the oral route; e) ability to read and comprehend any employed questionnaires/scales; f) signed informed consent;

Exclusion Criteria:

a) organic disease b)some other FGID (not IBS) or lactose intolerance c) having already followed an exclusion diet d)in case of pregnancy e)eating disorders f) prior surgery of the gastrointestinal tract g) neurodevelopmental disabilities

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | from running in and during all the dietetic treatment
  0-10
Irritable bowel Syndrome-Severity score | 15 days
  Is a five-item questionnaire measuring frequency and intensity of abdominal pain, the severity of abdominal distension, dissatisfaction with bowel habits, and the interference of IBS with daily life, scoring from 0 to 500. Cut-off of to evaluate the severity of IBS: < 175 for mild IBS, 175-300 for moderate IBS, and > 300 for severe IBS

SECONDARY OUTCOMES:
Fecal and urinary Metabolome | 14 days
  SCFA and VOCs

CONTACTS AND LOCATIONS:
Overall Officials: Ruggiero Francavilla, Prof, Principal Investigator — Interdisciplinary department of Medicine Pediatric section. University of Bari Aldo Moro
Locations (1):
- Pediatric Department "B Trambusti" Ospedale Giovanni XXIII Via Amendola 270, Bari, Ba, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and CSR will be available on request via email (fernandacristofori@gmail.com)
Supporting Information: Study Protocol, CSR
Time Frame: Available on request
Access Criteria: Request via email at fernandacristofori@gmail.com

REFERENCES:
- [Result] Caponio GR, Celano G, Calabrese FM, Riezzo G, Orlando A, D'Attoma B, Ignazzi A, Vacca M, Porrelli A, Tutino V, De Angelis M, Giannelli G, Russo F. Evaluation of the Effects of the Tritordeum-Based Diet Compared to the Low-FODMAPs Diet on the Fecal Metabolome of IBS-D Patients: A Preliminary Investigation. Nutrients. 2022 Nov 2;14(21):4628. doi: 10.3390/nu14214628. PMID 36364888
- [Result] Halmos EP, Christophersen CT, Bird AR, Shepherd SJ, Gibson PR, Muir JG. Diets that differ in their FODMAP content alter the colonic luminal microenvironment. Gut. 2015 Jan;64(1):93-100. doi: 10.1136/gutjnl-2014-307264. Epub 2014 Jul 12. PMID 25016597
- [Result] Staudacher HM, Lomer MCE, Farquharson FM, Louis P, Fava F, Franciosi E, Scholz M, Tuohy KM, Lindsay JO, Irving PM, Whelan K. A Diet Low in FODMAPs Reduces Symptoms in Patients With Irritable Bowel Syndrome and A Probiotic Restores Bifidobacterium Species: A Randomized Controlled Trial. Gastroenterology. 2017 Oct;153(4):936-947. doi: 10.1053/j.gastro.2017.06.010. Epub 2017 Jun 15. PMID 28625832
- [Result] Hyams JS, Di Lorenzo C, Saps M, Shulman RJ, Staiano A, van Tilburg M. Functional Disorders: Children and Adolescents. Gastroenterology. 2016 Feb 15:S0016-5085(16)00181-5. doi: 10.1053/j.gastro.2016.02.015. Online ahead of print. PMID 27144632